CLINICAL TRIAL: NCT05926193
Title: Arraigados Juntos - Rooted Together, Food as Medicine Project
Brief Title: Food as Medicine Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00111072
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Workshops (Experimental)
  Interventions: Dietary Supplement: Tailor Food Bags
- No Workshops (No Intervention)

INTERVENTIONS:
Dietary Supplement: Tailor Food Bags — The treatment group will participate in 6 nutrition workshops over the course of 6 months as well as receive weekly food bags that have been tailored for a DASH diet.
  Other Names: Nutrition Workshops
  Arms: Nutrition Workshops

SUMMARY:
Causes' Fresh Produce Program (FPP) in Durham County has addressed barriers to food security related to transportation with an innovative delivery model, but lacks evidence regarding the impact of food supplementation on chronic diseases like hypertension, which is prevalent in historically excluded populations in Durham County. The goal of this research study is to determine the efficacy of the modified Dietary Approach to Stop Hypertension (DASH) diet in Black/African American and Hispanic/Latinx participants with chronic hypertension who identify as food insecure using a randomized controlled trial. This research will leverage FPP's innovative distribution system to deliver medically-tailored produce bags and provide education workshops to the experimental participants relative to their experimental group. The study population group intends to include members of the Durham community and surrounding areas that identify as members of either the Black/African American or Hispanic/Latinx populations. Success will be measured in pre- and post-intervention biomarkers and qualitative participant experience data. Recognizing the risk of using Protected Health Information of Durham community members, many of whom are members of historically excluded populations that have been subjugated to harmful and extractive research practices, steps will be taken to ensure that collected information about research participants' personal and health information is protected and used only for the purposes of research. Ultimately, this research aims to work directly with the community to address hypertension outside of the clinic using food and education delivered directly to participants. The success of such an intervention could lead to expansion of delivering medically and culturally tailored foods to the larger FPP population and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. Adult parent/legal guardian (age 18 or older)
2. Documented essential hypertension (systolic BP >140 and/or diastolic BP >90, at least two documented clinical measurements)
3. Self-reported African American or Latino

Exclusion Criteria:

1. Hypertension due to secondary cause (e.g. renovascular hypertension, hyperthyroidism, Cushing's disease etc.)
2. Homelessness or insecure/transitional housing
3. Inability to prepare or cook food for themselves
4. Participants not living in Durham County, N.C.
5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 6 weeks, 12 weeks
  Systolic and diastolic BP will be documented at end of visit

SECONDARY OUTCOMES:
Patient satisfaction with culturally relevant foods | 12 weeks
  Survey/ Likert Scale 1- not satisfied- 5 Very Satisfied and open comments

OTHER OUTCOMES:
satisfaction with nutrition education sessions | 12 weeks
  Survey/ Likert Scale 1- not satisfied- 5 Very Satisfied and open comments
satisfaction with the DASH diet, | 12 weeks
  Survey/ Likert Scale 1- not satisfied- 5 Very Satisfied and open comments

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No